CLINICAL TRIAL: NCT04339803
Title: Dose-Finding of Lower Limb Mirror Therapy After Stroke.
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of East Anglia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 255913
Record Dates: First submitted 2020-03-23; First posted 2020-04-09 (Actual); Last update posted 2021-11-08 (Actual); Status verified 2021-11

CONDITIONS: Stroke
Keywords: Mirror therapy; Rehabilitation; Lower limb; Motor recovery
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- mirror therapy (Experimental): lower limb mirror therapy using ankle exercise
  Interventions: Other: rehabilitation intervention

INTERVENTIONS:
Other: rehabilitation intervention — we use lower limb mirror therapy after stroke for two weeks

SUMMARY:
This study will investigate the maximum dose per day of using mirror therapy for ankle exercise after stroke. The design is a 3+3 rule based, dose- finding study. Each cohort will consist of three participants. The first cohort will be assigned to do a dose of 15 minutes each day for two weeks. The second and subsequent cohorts will exercise at target dose set accordance to the nine preset rules and the modified Fibonacci sequence (mFBS).The study will continue until the stopping rule is triggered. The last dose tested will be identified as the maximum tolerable dose per day.

DETAILED DESCRIPTION:
Procedure:a 3+3 rule-based, dose-escalation design (Colucci et al,2017). recruitment process: the study will begin with a cohort of three participants (n=3). Each of the subsequent cohorts will also be of three participants. The start dose will be set at 15 minutes (cohort one). Participants will do ankle dorsiflexion exercise at the set dose with the mirror for two weeks. The second and subsequent cohorts will exercise at dose set in accordance to the nine preset rules and the modified Fibonacci sequence (mFBS) .

Sample size: The target sample size is not usually predefined for a dose-finding study. The final sample size will be determined by the response of consecutive cohorts to the set dose. Usually, in pharmaceutical dose-finding studies, the sample size lies between 12 and 40.

Data analysis : The data for each cohort will be analysed using descriptive statistics. No significance testing is involved.

ELIGIBILITY:
Inclusion Criteria:

* Participants have had a stroke for six weeks or more before recruitment to this study, and are discharged from NHS statutory stroke rehabilitation.
* Participants will be at least 18 years of age
* Able to produce some voluntary contraction of paretic ankle ( motricity index between 9 and 19).
* Ability to understand and follow simple verbal instructions (one-stage commands), i.e. sufficient communication, orientation, and memory to participate in mirror therapy ankle exercise.
* Participants will have had no lower limb injury in the last six months and were able to walk independently indoors before the index stroke.

Exclusion Criteria:

* Foot or ankle contracture that prevents 50% of the passive range of motion.
* Any condition that can be exaggerated by performing the therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2019-04-23 (Actual); Primary Completion 2021-08-09 (Actual); Study Completion 2021-08-09 (Actual)

PRIMARY OUTCOMES:
Changes in the Motricity Index | Baseline, 2 weeks.

SECONDARY OUTCOMES:
Changes in the Symmetry | Baseline, 2 weeks
  in Tibialis anterior muscle activation between the more and less paretic leg
Changes in the Neural excitability | Baseline, 2 weeks
  at the spinal level using peripheral nerve stimulation-H reflex
changes in the Transcranial magnetic stimulation (TMS) | Baseline, 2 weeks
  Corticospinal tract excitability

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Pomeroy, Professor, Study Director — School of Health Sciences, University of East Anglia
Locations (1):
- Sarah Bajuaifer, Norwich, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Participant data only will be shared with the research team

REFERENCES:
- [Derived] Bajuaifer S, Grey MJ, Hancock NJ, Chandler E, Pomeroy VM. Maximum tolerable daily dose of mirror movement therapy ankle exercises after stroke: an early phase dose screening study. Physiotherapy. 2024 Mar;122:30-39. doi: 10.1016/j.physio.2023.10.007. Epub 2023 Nov 4. PMID 38237263